CLINICAL TRIAL: NCT01551082
Title: Outpatient Chest Tube Management Following Thoracic Resection Improves Patient Length of Stay and Satisfaction Without Compromising Outcomes
Status: Terminated | Type: Observational
Why Stopped: Poor accrual
Sponsor: Alliance of Cardiothoracic and Vascular Surgeons (Other)
Responsible Party: Principal Investigator, Jeremy Smith, Registered Nurse, Alliance of Cardiothoracic and Vascular Surgeons
Other Study IDs: MEM Chest tube study
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer; Pneumothorax; Subcutaneous Emphysema
MeSH Terms: conditions — Lung Neoplasms; Pneumothorax; Subcutaneous Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Outpatient chest tubes: All patients, mixed gender, race, and age, who underwent thoracic resection by one surgeon over the past seven years and discharged home with air leak present and chest tube to portable drainage device.

SUMMARY:
Discharging patients home with air leak and chest tube to portable drainage device after thoracic resection is cost effective and safe without compromising patients outcome or satisfaction. Despite good outcomes this practice is not done universally by thoracic surgeons.

DETAILED DESCRIPTION:
Medical chart database to identify patients ,of one thoracic surgeon over the last seven years, who underwent thoracic resection and were discharged home with an air leak and chest tube to portable drainage device was completed. Once all patients were identified, all possible vulnerable patients were discarded. Written consent for participation was obtained by eligible patients and subjects willing to participate were given further explanation of the study. All willing participants completed an Outpatient Chest Tube Quality of Life Questionnaire. Upon completion of the questionnaire participants involvement in the study was complete. Data was collected and correlations between variables statistically analysed to determine significant factors affecting care.

ELIGIBILITY:
Inclusion Criteria:

* all patients 18-89,
* all genders,
* all patients undergoing thoracic resection,
* all patients discharged with chest tube

Exclusion Criteria:

* minors,
* all patients > 90 years old,
* all mentally challenged,
* all non-English speaking patients

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracic resection by one surgeon with post operative air leak being discharged home with chest tube and portable drainage device.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy S Smith, BSN, Principal Investigator — Alliance of Cardiac Thoracic and Vascular Surgeons
Locations (1):
- Memorial Hospital, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 years in medical clinic
Period: Overall Study
Arm/Group | Outpatient Chest Tubes
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patients older than 18 years old who underwent lung resection and were sent home with chest tubes
Arm/Group | Outpatient Chest Tubes
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — All patients > 18 years or older, mixed gender, race, and age who underwent thoracic resection by one surgeon and were discharged home with air leak present and chest tube to portable drainage device
  Participants
    <=18 years | 0
    Between 18 and 65 years | 4
    >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Outpatient Chest Tube Management Following Thoracic Resection Improves Patient Length of Stay and Satisfaction Without Compromising Outcomes
Description: Outcome measures for this study were to correlate outpatient chest tube management with patient satisfaction. Also to correlate decreased length of stay without compromising any patient outcomes.
Time Frame: 2 years
Population: Study was terminated and no data were collected for the outcome
Arm/Group | Outpatient Chest Tubes
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Outpatient Chest Tubes
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes